CLINICAL TRIAL: NCT05992181
Title: Development of a Digital Tool for the Individualization of Speech Therapy Care for Premature Newborns
Acronym: NEORTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A01290-45
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): With the speech therapy already in place in the department.
- experimental group (Experimental): With the speech therapy already in place in the department, plus access to videos and the introduction of early orofacial stimulation.
  Interventions: Other: NEORTHO

INTERVENTIONS:
Other: NEORTHO — early orofacial stimulation
  Arms: experimental group

SUMMARY:
The study concerns the creation and implementation of a digital tool presenting the various orofacial stimuli that can be offered to premature newborns. This app is intended for parents, to allow them to play a more active role in their child's care, and provide them with special time with their child. The notion of pleasure is very important to us, and it's vital to help parents rediscover this feeling with their child. Different profiles will be created to individualize our recommendations, facilitate the understanding of orofacial stimuli, make them more concrete than drawings, and provide care adapted to each patient and improve the development of newborns through more regular orofacial stimulation.

DETAILED DESCRIPTION:
Two groups will be formed:

Group A - control: receiving the speech therapy currently in place in the department.

Group B - experimental: will receive the same care as the first group, plus access to the videos and the introduction of early orofacial stimulation.

Group B: First, an initial assessment will be performed in speech-language pathology of the oro-myofunctional and oral functions of the newborn. This will determine which orofacial solicitations to give to the baby and create in the patient's profile.

Parents will be trained in orofacial stimulation and will be coached during the first sessions. When parents are ready, access will be given to their personal space on the application. Appointments will be scheduled to remodel the treatment if necessary. Sucking (ECEPAB), feeding (PIBBS) and behavioural (EDIN) abilities will be assessed. Parents will be asked to fill out a questionnaire about their feelings.

ELIGIBILITY:
Inclusion Criteria:

* Child born prematurely before 29 weeks of amenorrhea (SA).
* Alive for minimum 24h.
* Holders of parental authority who have been informed of the study and have not objected.

Exclusion Criteria:

* Child born after 29 weeks of amenorrhea.
* with a genetic or severe neurological pathology or withdrawal syndrome.
* with a vital prognosis.
* whose family home is too far from the service.

Ages: 24 Hours to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Milk taken daily | up to 3 months
  Percentage of the amount of milk taken daily (measure taken once per week throughout the study).

SECONDARY OUTCOMES:
Behavior scale for the analysis of oral reflexes and suction reflexes (MIAM questionnaire) | Day 0, Day 15, Day 30, Day 45, Day 60, Day 75, Day 90
  Analysis of oral and suction reflexes : global observation and functional assessment. (0=absent to 2=normal)
Feeding behavior scale for premature infants moving to bottle-feeding (ECEPAB questionnaire | Day 0, Day 15, Day 30, Day 45, Day 60, Day 75, Day 90
  feeding behavior scale for premature infants moving to bottle-feeding (0=absent to 18=normal)
Milk flower (PIBBS questionnaire) | Day 0, Day 15, Day 30, Day 45, Day 60, Day 75, Day 90
  global observation and functional assessment (0=absent to 20=normal)
Newborn Pain and Discomfort Scale (EDIN questionnaire) | Day 0, Day 15, Day 30, Day 45, Day 60, Day 75, Day 90
  Newborn Pain and Discomfort Scale (0=normal to 15=painful)
anxiety questionnaire | Day 0, Day 30, Day 60, Day 90
  anxiety questionnaire for the parents (0=relaxed to 2=anxious)
satisfaction questionnaire | Day 90
  satisfaction questionnaire for the application (0=unsatisfied to 3=satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No